CLINICAL TRIAL: NCT03256526
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, 3-ARM, PARALLEL- GROUP STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACODYNAMICS OF PF-06835919 ADMINISTERED ONCE DAILY FOR 6 WEEKS IN ADULTS WITH NONALCOHOLIC FATTY LIVER DISEASE
Brief Title: 6-week Safety and PD Study in Adults With NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C1061003
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Results first posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — PF-06835919

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06835919 Low Dose (Experimental): 75 mg once daily
  Interventions: Drug: PF-06835919 Low Dose
- PF-06835919 High Dose (Experimental): 300 mg once daily
  Interventions: Drug: PF-06835919 High Dose

INTERVENTIONS:
Drug: Placebo — 0 mg
  Arms: Placebo
Drug: PF-06835919 Low Dose — 75 mg once daily
  Arms: PF-06835919 Low Dose
Drug: PF-06835919 High Dose — 300 mg once daily
  Arms: PF-06835919 High Dose

SUMMARY:
IN THIS PHASE 2A, RANDOMIZED, DOUBLE BLIND, PLACEBO CONTROLLED, 3 ARM, PARALLEL- GROUP STUDY, SAFETY, TOLERABILITY, AND PHARMACODYNAMICS OF PF-06835919 ADMINISTERED ONCE DAILY FOR 6 WEEKS WILL BE ASSESSED IN ADULTS WITH NONALCOHOLIC FATTY LIVER DISEASE

ELIGIBILITY:
Inclusion Criteria:

* BMI at least 28 kg/m2
* Type 2 diabetes and/or metabolic syndrome

Exclusion Criteria:

* Liver disease
* Type 1 diabetes
* Recent heart attack or stroke
* Inability to have an MRI scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - National Research Institute, Los Angeles, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Stand-Up MRI of Miami, Miami, Florida
  - Avail Clinical Research, LLC, Orange City, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - WR-ClinSearch LLC, Chattanooga, Tennessee
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - National Clinical Research, Inc, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kazierad DJ, Chidsey K, Somayaji VR, Bergman AJ, Birnbaum MJ, Calle RA. Inhibition of ketohexokinase in adults with NAFLD reduces liver fat and inflammatory markers: A randomized phase 2 trial. Med. 2021 Jul 9;2(7):800-813.e3. doi: 10.1016/j.medj.2021.04.007. Epub 2021 Apr 27. PMID 35590219
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1061003&StudyName=A+Phase+2a%2C+Randomized%2C+Double-blind%2C+Placebo-controlled%2C+3-arm%2C+Parallel-+Group+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Pharmacodynamics+Of+Pf-06835919+Administered+Once+Daily+For+6+Weeks+In+Adults+With+Nonalcoholic+Fatty+Liver+Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-06835919 tablets once daily (QD) were administered orally.
- PF-06835919 75 mg: PF-06835919 75 mg tablets QD were administered orally.
- PF-06835919 300 mg: PF-06835919 300mg tablets QD were administered orally.
Period: Overall Study
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
Started | 19 | 17 | 17
Completed | 17 | 17 | 14
Not Completed | 2 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all eligible participants who received the study medication.
Groups:
- PF-06835919 300 mg: PF-06835919 300 mg tablets QD were administered orally.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg | Total
Number analyzed (Participants) | 19 | 17 | 17 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.00 (9.67) | 52.82 (8.17) | 52.29 (9.26) | 52.00 (8.94)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 6 | 2 | 3 | 11
  45-64 Years | 13 | 15 | 14 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 10 | 26
  Male | 12 | 8 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 6 | 10 | 31
  Not Hispanic or Latino | 4 | 11 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 10 | 12 | 39
  Black or African American | 2 | 6 | 5 | 13
  Asian | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
Age Range [Median (Full Range); unit: Years] | 53.00 [31 to 63] | 54.00 [32 to 64] | 54.00 [31 to 63] | 54.00 [31 to 64]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Whole Liver Fat at Week 6
Description: The percent change from baseline in whole liver fat at Week 6 was assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF).
  MRI-PDFF generates measures of the fraction of mobile protons in the liver attributable to fat content and provides whole liver coverage so that fat content can be assessed across 8 Couinaud liver segments. Whole liver PDFF was calculated as follows:
  Whole Liver PDFF= PDFFs for (Segment I+Segment II+Segment III+Segment IVa+Segment IVb+Segment V+Segment VI+Segment+VII+Segment VIII) / (number of segments assessed).
  The same segments were to be used at both baseline and post-baseline time points in the calculation of whole liver PDFF to derive the percent change from baseline.
  The values of whole liver PDFF ranges from 0 to 100 and higher values represent higher liver fat.
Time Frame: Baseline and Week 6
Population: The efficacy analysis population was defined as all randomized participants who received at least 1 dose of randomized treatment and assessed by MRI-PDFF at Week 6.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
Number analyzed (Participants) | 17 | 17 | 13
Percent Change | -7.97 (24.521) | 2.84 (22.246) | -25.43 (22.434)
Statistical Analysis 1: Comparison: Placebo vs PF-06835919 75 mg; Test type: Superiority; p = 0.1654, ANCOVA; LS mean difference = 11.45, 90% CI 2-sided [-2.19 to 25.09]
Statistical Analysis 2: Comparison: Placebo vs PF-06835919 300 mg; Test type: Superiority; p = 0.0395, ANCOVA; LS mean difference = -18.73, 90% CI 2-sided [-33.55 to -3.90]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: All-causality adverse events (AEs) were any untoward medical occurrence in a study participant who administered a product or medical device, the event need not necessarily have a causal relationship with the treatment or usage. Treatment-related AEs were any untoward medical occurrence in a study participant who administered a product or medical device, the event needed to have a causal relationship with the treatment or usage.
  A TEAE was defined as any event not present prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments.
Time Frame: Baseline up to Day 77 (28-35 days post last dose)
Population: The safety analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
Number analyzed (Participants) | 19 | 17 | 17
Participants
  All-causality TEAEs | 5 | 4 | 5
  Treatment-related TEAEs | 0 | 1 | 1

3. Secondary Outcome: Number of Participants With Post-dose Vital Signs Data Meeting Categorical Criteria
Description: The vital sign categorical criteria included:
  Sitting DBP (diastolic blood pressure) millimeter of mercury (mmHg) Change >= 20 mmHg increase Sitting SBP (systolic blood pressure) (mmHg) Change >= 30 mmHg increase Sitting DBP (mmHg) Change >= 20 mmHg decrease Sitting SBP (mmHg) Change >= 30 mmHg decrease Sitting DBP (mmHg) Value < 50 mmHg Sitting Pulse Rate (bpm) Value < 40 bpm or Value > 120 bpm Sitting SBP (mmHg) Value < 90 mmHg
Time Frame: Baseline up to Day 56 (Week 8)
Population: The analysis population included all participants who received at least 1 dose of investigational product and were evaluated against the criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
Number analyzed (Participants) | 18 | 17 | 17
Participants
  Sitting DBP (mmHg) Change >= 20 mmHg increase | 1 | 0 | 1
  Sitting SBP (mmHg) Change >= 30 mmHg increase | 0 | 0 | 2
  Sitting DBP (mmHg) Change >= 20 mmHg decrease | 1 | 1 | 0
  Sitting SBP (mmHg) Change >= 30 mmHg decrease | 0 | 1 | 2
  Sitting DBP (mmHg) Value <50 mmHg | 0 | 0 | 0
  Sitting Pulse Rate (bpm) Value < 40 bpm | 0 | 0 | 0
  Sitting Pulse Rate (bpm) Value > 120 bpm | 0 | 0 | 0
  Sitting SBP (mmHg) Value < 90 mmHg | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Post-dose ECG Data Meeting Categorical Criteria
Description: The ECG categorical criteria included:
  PR Interval (msec) percent (%)Change >= 25% increase when baseline >200 or >=50% increase when baseline <=200 QRS Interval (msec) %Change >= 50% increase QTcF Interval (Fridericia's Correction) (msec) increase 30 <= Change < 60 or Change >= 60 PR Interval (msec) Value >= 300 QRS Interval (msec) Value >= 140 QTcF Interval (Fridericia's Correction) (msec) 450 <= Value <480 or 480 <=Value <500 or Value >= 500
Time Frame: Baseline up to Day 56 (Week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
Number analyzed (Participants) | 18 | 17 | 17
Participants
  PR Interval (msec) %Change >= 25/50% increase | 0 | 0 | 0
  QRS Interval (msec) %Change >= 50% increase | 0 | 0 | 0
  QTcF Interval (msec) 30<= Change < 60 increase | 1 | 0 | 0
  QTcF Interval (msec) Change >= 60 increase | 0 | 0 | 0
  PR Interval (msec) Value >= 300 | 0 | 0 | 0
  QRS Interval (msec) Value >= 140 | 0 | 0 | 0
  QTcF Interval (msec) 450 <= Value <480 | 1 | 1 | 0
  QTcF Interval (msec) 480<= Value < 500 | 0 | 0 | 0
  QTcF Interval (msec) Value >= 500 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Below parameters were evaluated for laboratory tests: Hemoglobin, Hematocrit, Erythrocytes, Ery. Mean Copuscular Volume, Ery. Mean Copuscular Hemoglobin, Ery. Mean Corpuscular HGB Concentration, Platelets, Leukocytes, Lymphocytes, Neuprophils, Basophils, Eosinophils, Monocytes, Bilirubin, Direct Biliirubin, Indirect Bilirubin, Aspartate Aminotransferase, Alanine Aminotransferase, Gamma Glutamyl Transferase, Alkaline Phosphatase, Protein, Albumin, Albumin, Blood Urea Nitrogen, Creatinine, Urate, Sodium, Potassium, Chloride, Calcium, Bicarbonate, Glucose-Fasting, pH, Urine Glucose, Ketone, Urine Protein, Urine Hemoglobin, Urobilinogen, Urine Bilirubin, Nitrite, Leukocyte Esterase, Urine Erythocytes, Urine leukocytes, Hyaline Casts, Urine Creatinine.
Time Frame: Baseline up to Day 56 (Week 8)
Population: The analysis population included participants with at least 1 observation of the given laboratory test while on study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
Number analyzed (Participants) | 18 | 17 | 17
Participants | 9 | 8 | 8

ADVERSE EVENTS:
Time Frame: Baseline up to Day 77 (28-35 days post last dose)
Arm/Group | Placebo | PF-06835919 75 mg | PF-06835919 300 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 5/19 | 4/17 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | PF-06835919 75 mg (N=17) | PF-06835919 300 mg (N=17)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclosure previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03256526/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT03256526/SAP_001.pdf